CLINICAL TRIAL: NCT04678232
Title: Treatment of Stress-Related Psychopathology: Targeting Maladaptive and Adaptive Event Processing
Brief Title: Positive Processes and Transition to Health
Acronym: PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University of Washington (Other); University of Delaware (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Norah Feeny, Professor, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R61MH113646; 5R61MH118401-02 (NIH)
Record Dates: First submitted 2020-12-08; First posted 2020-12-21 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder; Post Traumatic Stress Disorder
Keywords: transdiagnostic intervention; ptsd; posttraumatic stress disorder; mdd; major depressive disorder; adult; therapy; mental health; destabilizing life events; stressful life events
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: All participants will receive PATH therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- receive PATH therapy (Experimental): PATH includes six 60-90 min, weekly sessions, with two booster sessions for partial responders. Session 1 provides the PATH rationale and a review of life events (PATH of life: negative and positive). A rationale for an explicit focus on positive events/emotions will be provided. Sessions 2-4 focus on a verbal narrative of the destabilizing life event, reminiscence and processing of a major positive life event, and real-life practice to enact what was taught. Sessions 5 focuses on constructive processing and provides opportunity for integration and consolidation of learning. Session 6 focuses on future negative and positive events to promote application of new learning and resilience. Booster sessions focus on positive and negative life events since the last session and adaptive processes (constructive processing, approach, and reward). All sessions will include cultivation and elaboration of positive emotions to promote engagement and to build on the benefits of positive emotions.
  Interventions: Behavioral: Positive Processes and Transition to Health (PATH)

INTERVENTIONS:
Behavioral: Positive Processes and Transition to Health (PATH) — See arm/group description for details regarding this intervention
  Other Names: PATH

SUMMARY:
The R61 will be an open trial to determine if Positive Processes and Transition to Health (PATH) engages the proposed targets: unproductive processing, avoidance, and reward deficits in a sample of 45 adults who have experienced a destabilizing life event involving profound loss or threat, report persistent stressor-related symptoms of PTSD and/or depression, and are elevated on symptoms related to 2 of the 3 therapeutic targets. Additionally, will examine whether patients perceive PATH as helpful and complete/adhere to treatment, and therapist fidelity. Patients will receive 6 sessions of PATH (with 2 boosters, if partial responders). Primary targets will be assessed at pre-treatment, week 4, post-treatment, and at 1- and 3-month follow-up; secondary targets at pre-treatment, weekly during treatment, post-treatment, and at 1- and 3-month follow-ups.

DETAILED DESCRIPTION:
Evidence-based psychotherapies for posttraumatic stress disorder (PTSD) and depression consistently produce strong, clinically meaningful effects for many individuals. However, these interventions also have significant dropout rates, a large minority of individuals continue to have debilitating symptoms, and even those who respond may be vulnerable to relapse upon future stressors. More efficient and mechanistically precise interventions are needed. Consistent with the cross-cutting theme of studying the role of the environment in the NIMH Strategic Plan, the etiological role of exposure to destabilizing, stressful life events is common to both PTSD and depression. Not only do they share common distress-related triggers, symptoms, and maintaining processes, but they also commonly co-occur (upwards of 60%). Current PTSD and depression treatments typically focus on their respective disorders rather than on common processes that maintain psychopathology; and, importantly, they do not explicitly target positive adaptive processes associated with resilience. Decades of experimental studies, prospective studies, and psychotherapy trials have identified interconnected maladaptive and adaptive processes associated with persistent psychopathology after stressful, destabilizing events. These maladaptive processes include: 1) unproductive event processing; 2) avoidance; and 3) reward sensitivity and processing deficits. These processes prolong negative mood, interfere with adaptive coping and processing of emotional material, and increase sensitivity to future stressful life events. PATH (Positive Processes and Transition to Health) directly targets these maladaptive processes while also teaching parallel adaptive skills (constructive processing, approach, and positive emotion processing and reward seeking). Six, 90-min sessions target individuals who have experienced a destabilizing life event and have persistent stressor-related symptoms. PATH utilizes life event processing (revisiting, meaning making), focusing repeatedly on an identified destabilizing life event, positive life events, and future events as a framework to identify maladaptive processes and teach constructive processing skills. PATH has the potential to reduce dropout, improve treatment engagement and outcomes, identify potential treatment mechanisms, and ultimately reduce the costly human and economic burden of stressor-related psychopathology.

For the open trial's "Go" to be achieved and to proceed to the R33, two criteria must be met. The first is that at least 2 of the 3 primary targets must change via PATH. A moderate effect size (d = 0.60) was chosen to reflect evidence of clinically meaningful target engagement (see Gold et al., 2017), in line with NIMH guidelines for a preliminary signal of target engagement/efficacy in intervention trials. Second, at least one of the secondary measures must show a moderate effect (d = 0.50) from pre- to post-treatment. We included measures of each of the targets, as they are conceptualized as interrelated parts of a "stuck" system. For "Go" to an R01 after the R33, in addition to target engagement, primary outcomes of PTSD and depression must show clinically meaningful gains (e.g., Barth et al., 2016; Cusak et al., 2016).

ELIGIBILITY:
Inclusion Criteria:

* Destabilizing life event involving profound loss or threat, with a minimum duration of 12 weeks since the event, but occurred within the last 5 years.
* Between the ages of 18 and 65.
* Elevated target: Scores of at least moderate (1 or higher) on at least 2 of the 3 target mechanisms: re- experiencing or ruminative processing of the destabilizing event (PSS-I items: 1, 2, 3, 4 or QIDS-C item 11), avoidance (PSS-I items 6, 7, 8), or reward deficits (PSS-I items 12, 13, or QIDS-C item 13).

Exclusion Criteria:

* Current diagnosis of schizophrenia, delusional disorder, or organic mental disorder as defined by DSM-5.
* Current diagnosis of bipolar disorder, depression with psychotic features, or depression severe enough to require immediate psychiatric treatment (i.e., serious suicide risk with intent and plan).
* Severe self-injurious behavior or suicide attempt within the previous three months.
* Unwilling or unable to discontinue current cognitive behavioral psychotherapy.
* No clear memory of the destabilizing event or event occurred before age 3.
* Unstable dose of psychotropic medications in prior 3 months.
* Ongoing intimate relationship with the perpetrator (in assault related event).
* Current diagnosis of a substance use disorder (DSM-5).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norah C Feeny, PhD, Principal Investigator — Case Western Reserve University
Locations (3):
- United States (3):
  - University of Delaware, Newark, Delaware
  - Case Western Reserve University, Cleveland, Ohio
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Receive PATH Therapy
Started | 45
Completed | 40
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Receive PATH Therapy
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.98 (14.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 35
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 45
Affective Updating Task [Mean (Standard Deviation); unit: units on a scale] — The Affective Updating task (Pe et al., 2013; Pe, Raes, et al., 2013) measures updating of affective information in working memory. The task requires participants to continuously monitor and modify relevant affective information in working memory. Performance is inhibited by rumination. Forty-seven positive and 49 negative words are included. The AUT is scored using the mean proportion of correct responses. Scores for the AUT range from 0 to 1. Lower scores reflect greater deficits in affecting updating, while higher scores indicate greater abilities with affective updating.
  units on a scale | 0.38 (0.23)
Idiographic Behavioral Approach Task [Mean (Standard Deviation); unit: units on a scale] — The Idiographic Behavioral Approach Task (BAT; Mori & Aermendariz, 2001; Haynes, 2001) will use in vivo confrontation with feared or avoided stimuli measuring avoidance behavior. The task requires participants to rate their subjective units of distress (SUDs) on a scale of 0-100 (0 = no distress, 100 = extreme distress). The primary outcome measured is mean peak SUDs across all items. Higher scores indicate a higher average level of distress across all items, and lower scores indicate less distress on average across all items.
  units on a scale | 55.00 (23.27)
Probabilistic Reward Task [Mean (Standard Deviation); unit: units on a scale] — The Probabilistic Reward Task (PRT) assesses reward responsivity (e.g., Der-Avakian et al. 2013; Pizzagalli et al., 2005, 2008, 2008). In each trial, participants choose which of 2 difficult-to-differentiate stimuli was presented. Correct identification of the "rich stimulus" is rewarded 3 times more frequently. Reward propensity is calculated by increase in response bias, which is a robust measure of reward sensitivity (Pizzagalli et al., 2005, 2008; Vrieze et al., 2013). PRT scores range between -.75 to .65 (-.75 = lower reward sensitivity, .65 = greater reward sensitivity).
  units on a scale | -0.08 (0.29)
Posttraumatic Cognitions Inventory [Mean (Standard Deviation); unit: units on a scale] — The Posttraumatic Cognitions Inventory (PTCI; Foa et al., 1999) is a self-report that measures negative posttraumatic stressor-related thoughts that can contribute to the development and maintenance of PTSD. The measure includes 33 items, which are measured on a scale from 1-7 with 1 indicating "totally disagree" and 7 indicating "totally agree." The total score for the PTCI ranges from 33 to 231 and is determined by summing the scores of each subscale. Higher scores reflect more rigid negative cognitions. Total scores were used. Population: Missing data
  units on a scale
    number analyzed (Participants) | 40
    (all) | 151.03 (42.07)
Behavioral Activation for Depression Scale [Mean (Standard Deviation); unit: units on a scale] — Behavioral Activation for Depression Scale (Secondary Measure; BADS; Kanter et al., 2006) is a 25- item self-report of approach and avoidance in cognitive and behavioral domains not specific to depression. Items are rated from 0 = Not at all to 6 = Completely. The measure contains four subscales which include Activation, Avoidance/Rumination, Work/School Impairment, and Social Impairment. Total scores, which range from 0-150 are calculated by summing the four subscales. A higher score indicates higher behavioral activation and lower scores indicate more depressive symptoms. Population: Missing data
  units on a scale
    number analyzed (Participants) | 40
    (all) | 71.35 (24.96)
Snaith-Hamilton Pleasure Scale [Mean (Standard Deviation); unit: units on a scale] — Snaith-Hamilton Pleasure Scale (SHAPS; Snaith et al., 1995). The SHAPS is a 14- item self-report measuring the capacity to experience pleasure. On a four-point scale (1 = Strongly Agree to 4 = Strongly Disagree), varying statements are rated (e.g., "I would find pleasure in small things"; "I would find pleasure in a telephone call from a friend"). The measure reflects a unidimensional construct of anhedonia (Leventhal et al., 2006; Nakonezny et al., 2010). Total scores are measured on a scale from 14 to 56 (14 = severe anhedonia, 56 = no anhedonia). Population: Missing data
  units on a scale
    number analyzed (Participants) | 40
    (all) | 25.25 (2.29)

OUTCOME MEASURES:

1. Primary Outcome: Affective Updating Task (Pe et al., 2013; Pe, Raes, et al., 2013)
Description: The Affective Updating task (Pe et al., 2013; Pe, Raes, et al., 2013) measures updating of affective information in working memory. The task requires participants to continuously monitor and modify relevant affective information in working memory. Performance is inhibited by rumination. Forty-seven positive and 49 negative words are included. Under high levels of stress, deficits in affective updating predict more depressive symptoms over one year (Pe et al., 2016) and efficiency of reappraisal (Pe et al., 2013). Affective updating in contrast, predicts subjective well-being (Pe et al., 2013). The AUT is scored using the mean proportion of correct responses across 4 types of stimulus sets (positive-positive-positive words, negative-negative-negative, positive-negative-positive, negative-positive-negative). Scores for the AUT range from 0 to 1. Lower scores reflect greater deficits in affecting updating, while higher scores indicate greater abilities with affective updating.
Time Frame: Score at 6 weeks (immediately post treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Receive PATH Therapy
Number analyzed (Participants) | 40
units on a scale | 0.54 (0.23)

2. Primary Outcome: Idiographic Behavioral Approach Task
Description: The Idiographic Behavioral Approach Task (BAT; Mori & Aermendariz, 2001; Haynes, 2001) will use in vivo confrontation with feared or avoided stimuli measuring avoidance behavior. Each BAT is unique to each participant (e.g., news/videos of similar events, pictures of loved one). A general list of idiographic stimuli will be developed with participants, who will then approach the stimuli.
  The task requires participants to rate their subjective units of distress (SUDs) on a scale of 0-100 (0 = no distress, 100 = extreme distress). The primary outcome measured is mean peak SUDs. The mean peak SUDs is calculated by averaging together all of the participant's reported SUDs measured at their highest level of distress. Higher scores indicate a higher average level of distress across all items, and lower scores indicate less distress on average across all items.
Time Frame: Score at 6 weeks (immediately post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Receive PATH Therapy
Number analyzed (Participants) | 37
score on a scale | 25.65 (22.47)

3. Primary Outcome: Probabilistic Reward Task (Pizzagalli et al., 2005)
Description: The Probabilistic Reward Task (PRT) assesses reward responsivity (e.g., Der-Avakian et al. 2013; Pizzagalli et al., 2005, 2008, 2008). In each trial, participants choose which of 2 difficult-to-differentiate stimuli was presented. Stimuli are groups of bunnies or dogs (diameter: 25 mm; eyes: 7 mm). Unknown to them, correct identification of the "rich stimulus" is rewarded 3 times more frequently ("Correct! You won 20 cents"). Reward propensity is calculated by increase in response bias during the final block relative to the first. Degree of response bias toward the frequently reinforced alternative is a robust measure of reward sensitivity (Pizzagalli et al., 2005, 2008; Vrieze et al., 2013). The PRT is administered online through Inquisit Lab on Millisecond. PRT scores range between -.75 to .65 (-.75 = lower reward sensitivity, .65 = greater reward sensitivity).
Time Frame: Score at 6 weeks (immediately post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Receive PATH Therapy
Number analyzed (Participants) | 40
score on a scale | -.03 (.25)

4. Secondary Outcome: Posttraumatic Cognitions Inventory (Foa et al., 1999)
Description: The Posttraumatic Cognitions Inventory (PTCI; Foa et al., 1999) is a self-report that measures negative posttraumatic stressor-related thoughts that can contribute to the development and maintenance of PTSD. The measure includes 33 items grouped into three subscales. The 21-item Negative Cognitions about Self scale measures negative self-perception since the traumatic event. The 7-item Negative Cognitions about the World subscale evaluates mistrust of others and perceptions of danger. The 5-item Self Blame scale measures self-blame since the traumatic incident. All items are measured on a scale from 1-7 with 1 indicating "totally disagree" and 7 indicating "totally agree." The total score for the PTCI ranges from 33 to 231 and is determined by summing the scores of each subscale. Higher scores reflect more rigid negative cognitions. Total scores were used.
Time Frame: Score at 6 weeks (immediately post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Receive PATH Therapy
Number analyzed (Participants) | 38
score on a scale | 102.05 (43.14)

5. Secondary Outcome: Behavioral Activation for Depression Scale (Kanter et al., 2006)
Description: Behavioral Activation for Depression Scale (Secondary Measure; BADS; Kanter et al., 2006) is a 25- item self-report of approach and avoidance in cognitive and behavioral domains not specific to depression. Items are rated from 0 = Not at all to 6 = Completely. The measure contains four subscales which include Activation, Avoidance/Rumination, Work/School Impairment, and Social Impairment. Total scores, which range from 0-150 are calculated by summing the four subscales. A higher score indicates higher behavioral activation and lower scores indicate more depressive symptoms. The BADS has good factor structure, internal consistency, construct, and predictive validity (Kanter et al., 2009; Manos et al, 2011) and sensitivity to change (d =.86; CBT for depression, O'Mahen et al., 2017).
Time Frame: Score at 6 weeks (immediately post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Receive PATH Therapy
Number analyzed (Participants) | 38
score on a scale | 106.5 (24.97)

6. Secondary Outcome: Snaith-Hamilton Pleasure Scale (Snaith et al., 1995)
Description: Snaith-Hamilton Pleasure Scale (SHAPS; Snaith et al., 1995). The SHAPS is a 14- item self-report measuring the capacity to experience pleasure. On a four-point scale (1 = Strongly Agree to 4 = Strongly Disagree), varying statements are rated (e.g., "I would find pleasure in small things"; "I would find pleasure in a telephone call from a friend"). The measure has good convergent and discriminant validity and reflects a unidimensional construct of anhedonia (Leventhal et al., 2006; Nakonezny et al., 2010). Total scores are measured on a scale from 14 to 56 (14 = severe anhedonia, 56 = no anhedonia).
Time Frame: Score at 6 weeks (immediately post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Receive PATH Therapy
Number analyzed (Participants) | 38
score on a scale | 21.79 (2.69)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from start of study procedures (e.g., enrollment) through 3 months post study completion (up to 6 months from study enrollment).
Arm/Group | Receive PATH Therapy
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT04678232/Prot_SAP_000.pdf